CLINICAL TRIAL: NCT04239404
Title: The Prognostic Impact of Periprocedural Myocardial Injury in Stable Coronary Artery Disease Patients Undergoing Elective Percutaneous Coronary Intervention
Brief Title: Prognostic Impact of PMI in Stable CAD Undergoing PCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PMI-CAD-PCI
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Periprocedural Myocardial Injury; Coronary Artery Disease; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples of the participants before and after percutaneous coronary intervention therapy were selected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PMI
- non-PMI

SUMMARY:
This is a single-center, observational, prospective study. This study aims to observe the effect of periprocedural myocardial injury on cardiovascular events in patients undergoing elective percutaneous coronary intervention, and to detect the levels of serum inflammatory factors before and after intervention to predict the occurrence of periprocedural myocardial injury and its association with cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* underwent elective coronary stenting
* patients permit informed consents

Exclusion Criteria:

* acute STEMI
* NYHA class III-IV heart failure
* moderate-to-severe valvular disease
* missing post-PCI troponin results
* active infection, respiratory failure
* liver dysfunction (liver enzyme >3xURL or bilirubin >2xURL),
* malignancy and systemic connective tissue disease
* unable to get a informed consents

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-patients with stable coronary artery disease undergoing elective percutaneous coronary intervention in Zhongshan Hospital will be enrolled.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Major cardiac events | 12 months after PCI
  cardiac death, target vessel revascularization, target lesion revascularization, non-fatal myocardial infarction, heart failure, angina pectoris

SECONDARY OUTCOMES:
Serum level of inflammatory factors | 1 day after PCI
  Serum level of inflammatory factors including TNFα, IL-6 and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No